CLINICAL TRIAL: NCT03158480
Title: Safety and Efficacy of Immune Therapy for Condyloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20173357201827
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-03

CONDITIONS: Condylomata Acuminata
Keywords: DC-CIK; interferon
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DC-CIK+interferon Group (Experimental): dendritic cell-activated cytokine-induced killer cells (DC-CIK) immunotherapy plus interferon intervention
  Interventions: Biological: DC-CIK immunotherapy
- Placebo+interferon Group (Placebo Comparator): saline as placebo plus interferon intervention
  Interventions: Biological: DC-CIK immunotherapy

INTERVENTIONS:
Biological: DC-CIK immunotherapy — Cytokine-induced killer (CIK) cells are co-cultured with HPV induced dendritic cells (DCs); HPV specific DC-CIK will be induced to condylomata acuminata patients

SUMMARY:
Cytokine-induced killer (CIK) cells will be co-cultured with HPV induced dendritic cells (DCs); HPV specific DC-CIK will be induced to Condylomata Acuminata patients using interferon, whose recurrence rate and total cost will be compared to Condylomata Acuminata patients only use interferon.

ELIGIBILITY:
Inclusion Criteria:All patients have typical clinical characters of condyloma, positive for HPV-DNA test; All patients have been treated for cryotherapy or laser plus interferon for over half a year without completely recovery. All patients or their family will sign informed consent and approved by Ethics Committee of Shenzhen Second People's Hospital -

Exclusion Criteria:pregnant, blood disease, contraindication for immune therapy, allergic to interferon

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-25 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Condylomata Acuminata recurrence rate | 6 months
  Condylomata Acuminata recurrence rate in 6 months after treatment

SECONDARY OUTCOMES:
skin tissue HPV gene | 6 months
  use PCR to testify skin tissue HPV gene
side effect | 6 months
  evaluate and record side effect of each group

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided